CLINICAL TRIAL: NCT06472167
Title: Impact of Breathing Exercises on Lung Function in Chronic Airway Diseases
Brief Title: Breathing Exercises on Lung Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Abd Elmoniem Mohamed, Lecturer of chest medicine, Mansoura University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R.24.05.2638
Record Dates: First submitted 2024-06-13; First posted 2024-06-25 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Breathing Exercises
Keywords: Breathing exercises; lung function; Chronic airway diseases
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic airway diseases treated by medication (No Intervention): Chronic airway diseases treated by medication without breathing exercises
- Chronic airway diseases treated by medication with breathing exercises (Active Comparator): Chronic airway diseases treated by medication and breathing exercises
  Interventions: Behavioral: Breathing exercises

INTERVENTIONS:
Behavioral: Breathing exercises — Breathing exercises as diaphragmatic breathing exercises and pursued lip breathing and incentive spirometry
  Other Names: Diaphragmatic Breathing exercise; Pursued lip breathing
  Arms: Chronic airway diseases treated by medication with breathing exercises

SUMMARY:
aim of this study is to evaluate the efficacy of pulmonary rehabilitation program as a non-pharmacological treatment method to: Improve functional capacity as assessed by six-minute walking distance (6MWD) test. Improve dyspnea level as assessed by Medical Research Council (MRC) dyspnea scale. Improve pulmonary function tests and arterial blood gas.

DETAILED DESCRIPTION:
Breathing exercises offer numerous benefits for individuals with chronic airway diseases, such as chronic obstructive pulmonary disease (COPD), asthma and bronchiectasis. These exercises help improve respiratory function, reduce symptoms, and enhance the overall quality of life.Techniques such as diaphragmatic breathing, incentive spirometer and pursed lip breathing help patients use their lungs more effectively. Breathing exercises can enhance lung function by increasing the efficiency of the respiratory muscles and improving ventilation. Asthma is a chronic inflammatory disorder of the airways classified as intermittent or persistent (mild, moderate or severe), according to the presence of diurnal and nocturnal symptoms, necessity of medication, frequency of exacerbation, physical activity limitations and pulmonary function. All of these symptoms deteriorate in the patient's quality of life and psychological well-being and restrict daily living physical activities (DLPA). Asthma symptoms experienced during daily living physical activities (DLPA) or the fear of triggering symptoms may keep asthmatic subjects from engaging in physical exercise, and the patients tend to be less physically active and less conditioned than healthy individuals. In addition, asthmatic patients have higher levels of anxiety and depression that have been shown to be associated with an increased number of exacerbations and the diagnosis of severe asthma. These psychosocial disorders can modify the respiratory breathing pattern, which leads to irregular breathing, frequent sighing, and predominant thoracic breathing. These irregular breathing patterns increase the number of respiratory (breathlessness, chest tightness and pain) and non-respiratory symptoms (anxiety, dizziness and fatigue). Recent Global Initiative for Chronic Obstructive Pulmonary Disease guidelines (GOLD) underline the importance of pulmonary rehabilitation (PR) as a part of an integrative multidisciplinary approach regardless of the stage of disease

ELIGIBILITY:
Inclusion Criteria:

* The patients fulfilled the criteria for COPD: the presence of a post bronchodilator FEV1 < 80% predicated together with an FEV1/FVC <0.70confirm the presence of airflow limitation that is not fully reversible.
* COPD patients ranging from mild to severe according to GOLD [stages I-IV].
* Asthmatic patients receive medical treatment for at least 6 months; and clinically stable (i.e., no exacerbation or changes in medication for ≥30 days).
* None of the individuals had been engaged in any exercise-training program before participating in the study.
* Optimized medical therapy according to GOLD & Global Initiative for Asthma (GINA)
* Clinically stable COPD and asthmatic patients (not suffering from a recent respiratory tract infection).
* All patients are Ex-smoker

Exclusion Criteria:

* Age <18 years.
* Pregnancy
* Current Smokers
* Patients that are incapable of exercising; unable to understand any questionnaire
* Multiple co- morbidity (e.g., cardiovascular diseases, active cancer)
* Neuromuscular disease as Myasthenia gravis, kypho-scoliosis
* Diaphragmatic Paralysis (paralyzed diaphragm exhibiting abnormal paradoxical movement, i.e., moving in a cranial direction during inspiration).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-08-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Impact of breathing exercises on Forced expiratory volume on first second (FEV1) in liter | 6 months
  Effect of Breathing exercises on lung function using spirometry
Impact of breathing exercises on Forced vital capacity (FVC) in liter | 6 months
  Effect of Breathing exercises on lung function using spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AbdElmoniem, Principal Investigator — Lecturer of chest medicine faculty of medicine Mansoura university
Locations (1):
- Mohamed AbdElmoniem, Al Mansurah, Egypt